CLINICAL TRIAL: NCT01577758
Title: An Open-Label, Dose Escalation, Phase 1, First-in-Human Study of MLN0264 in Adult Patients With Advanced Gastrointestinal Malignancies Expressing Guanylyl Cyclase C
Brief Title: Phase 1 Study of MLN0264 in Adult Patients With Advanced Gastrointestinal Malignancies Expressing Guanylyl Cyclase C
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C26001; 2011-002260-24 (EudraCT Number); U1111-1163-9720 (Registry Identifier: WHO)
Record Dates: First submitted 2012-04-02; First posted 2012-04-16 (Estimated); Results first posted 2016-07-25 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-09

CONDITIONS: Advanced Gastrointestinal Malignancies
Keywords: Phase 1,; Advanced gastrointestinal malignancies,; MLN0264,; Guanylyl Cyclase C(GCC),; Antibody Drug Conjugate(ADC)
MeSH Terms: interventions — indusatumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MLN0264 (Experimental): MLN0264 starting dose 0.3 mg/kg escalated until Maximum Tolerated Dose (MTD) was determined, 30-minute infusion, on Day 1 of each 21-Day treatment cycle.
  Interventions: Drug: MLN0264

INTERVENTIONS:
Drug: MLN0264 — MLN0264 30-minute infusion on Day 1 of each treatment cycle

SUMMARY:
This is an Open-Label, Multicenter, Dose Escalation, First-in-Human Study of MLN0264 in Adult Patients With Advanced Gastrointestinal Malignancies Expressing Guanylyl Cyclase C.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary consent form
* Diagnosis of GI malignancy with a GCC protein expressing tumor
* Male or female patients 18 years or older with measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST)
* Female patients who are post menopausal, surgically sterile, or agree to practice 2 effective methods of contraception or agree to abstain from heterosexual intercourse
* Male patients who agree to practice effective barrier contraception or agree to abstain from heterosexual intercourse
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Adequate bone marrow, hepatic and renal function as specified in the protocol

Exclusion Criteria:

* Female patients who are lactating or have a positive serum pregnancy test during the screening period
* Any serious medical or psychiatric illness that could interfere with the completion of treatment
* Major surgery or treatment with investigational drug before the first dose
* Serious infection within 14 days before the first dose of study drug
* Known HIV, inflammatory bowel disease, viral hepatitis or cerebral/meningeal brain metastases
* Patients with cardiovascular conditions specified in protocols
* Patients with history of another primary malignancy not in remission for at least 3 years

Please note that there are additional inclusion and exclusion criteria. The study center will determine if you meet all of the criteria.

Site personnel will explain the trial in detail and answer any question you may have if you do qualify for the study. You can then decide whether or not you wish to participate. If you do not qualify for the trial, site personnel will explain the reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2012-06; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Millennium Pharmaceuticals, Inc.
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 4 investigative sites in the United States and Spain from 11 June 2012 to 12 February 2014.
Pre-assignment Details: Participants with Gastrointestinal malignancies expressing guanylyl cyclase C were enrolled in the dose escalation phase: 0.3, 0.6, 1.2, 1.5, 1.8, 2.1 and 2.4 mg/kg to determine the maximum tolerated dose (MTD). MTD was established and participants were enrolled in the mCRC expansion phase. 3 participants were in both the 1.8 mg/kg and mCRC arms.
Groups:
- MLN0264 0.3 mg/kg: MLN0264 0.3 mg/kg, 30-minute intravenous (IV) infusion, Day 1 of each 21-day cycle, until disease progression or unacceptable toxicity or up to 1 year.
- MLN0264 0.6 mg/kg: MLN0264 0.6 mg/kg, 30-minute intravenous IV infusion, Day 1 of each 21-day cycle, until disease progression or unacceptable toxicity or up to 1 year.
- MLN0264 1.2 mg/kg: MLN0264 1.2 mg/kg, 30-minute intravenous (IV) infusion, Day 1 of each 21-day cycle, until disease progression or unacceptable toxicity or up to 1 year.
- MLN0264 1.5 mg/kg: MLN0264 1.5 mg/kg, 30-minute intravenous IV infusion, Day 1 of each 21-day cycle, until disease progression or unacceptable toxicity or up to 1 year.
- MLN0264 1.8 mg/kg: MLN0264 1.8 mg/kg, 30-minute IV infusion, Day 1 of each 21-day cycle, until disease progression or unacceptable toxicity or up to 1 year.
- MLN0264 2.1 mg/kg: MLN0264 2.1 mg/kg, 30-minute IV infusion, Day 1 of each 21-day cycle, until disease progression or unacceptable toxicity or up to 1 year.
- MLN0264 2.4 mg/kg: MLN0264 2.4 mg/kg, 30-minute IV infusion, Day 1 of each 21-day cycle, until disease progression or unacceptable toxicity or up to 1 year.
- MLN0264 1.8 mg/kg (mCRC Expansion): MLN0264 1.8 mg/kg, 30-minute IV infusion, Day 1 of each 21-day cycle, until disease progression or unacceptable toxicity or up to 1 year in participants with metastatic colorectal (rectal, colon, or colorectal) cancer (mCRC).
Period: Dose Escalation Phase
Arm/Group | MLN0264 0.3 mg/kg | MLN0264 0.6 mg/kg | MLN0264 1.2 mg/kg | MLN0264 1.5 mg/kg | MLN0264 1.8 mg/kg | MLN0264 2.1 mg/kg | MLN0264 2.4 mg/kg | MLN0264 1.8 mg/kg (mCRC Expansion)
Started | 2 | 2 | 2 | 2 | 6 | 4 | 1 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 2 | 2 | 2 | 2 | 6 | 4 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Not completed — Symptomatic Deterioration | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Progression Disease | 2 | 2 | 1 | 2 | 5 | 0 | 0 | 0
Period: mCRC Expansion Phase
Arm/Group | MLN0264 0.3 mg/kg | MLN0264 0.6 mg/kg | MLN0264 1.2 mg/kg | MLN0264 1.5 mg/kg | MLN0264 1.8 mg/kg | MLN0264 2.1 mg/kg | MLN0264 2.4 mg/kg | MLN0264 1.8 mg/kg (mCRC Expansion)
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 25
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 25
Not completed — Symptomatic Deterioration | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Progression Disease | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 19

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received at least 1 dose of study drug. A total of 41 participants participated in the study. There were 3 participants who participated in both phases of the study and are only counted once.
Groups:
- All Participants: All participants who participated in the Dose Escalation and mCRC Expansion Phases.
Arm/Group | All Participants
Number analyzed (Participants) | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.7 (10.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 27
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 34
  Not Reported | 2
Race/Ethnicity, Customized [Number; unit: participants]
  White | 39
  Not Reported | 2
Height [Mean (Standard Deviation); unit: cm] — Height data is only available for 39 participants.
  cm | 170.4 (7.69)
Weight [Mean (Standard Deviation); unit: kg] | 78.50 (18.573)
Body Surface Area [Mean (Standard Deviation); unit: m^2] — Body surface area data is only available for 39 participants.
  m^2 | 1.929 (0.2424)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-Limiting Toxicities (DLTs)
Description: DLT was defined as any of the following Adverse Events (AEs) that occur and are considered by the investigator to be related to therapy.
  1. Grade 4 neutropenia (Absolute Neutrophil Count < 500 cells/mm^3).
  2. Grade 3 or greater neutropenia with fever and/or infection.
  3. Grade 4 thrombocytopenia (platelets < 25,000/mm^3).
  4. Grade 3 or greater thrombocytopenia with clinically meaningful bleeding at any time.
  5. Grade 3 or greater nausea and/or emesis that occurs despite of prophylaxis.
  6. Grade 3 or greater diarrhea that occurs despite supportive care.
  7. Any other Grade 3 or greater non-hematological toxicity other than Grade 3 fatigue or Grade 3 Alopecia.
  8. Inability to start the next cycle of therapy due to treatment delay of more than 2 weeks because of lack of recovery.
  9. Other MLN0264-related non-hematologic toxicities Grade 2 or greater requiring discontinuation of therapy.
Time Frame: From the time informed consent is signed through 30 days after the last dose of study drug, approximately 9 months
Population: DLT evaluable Population: participants enrolled in the Dose Escalation phase of the study who either experienced a DLT during Cycle 1 or received a scheduled Cycle 1 dose and completed all study procedures in Cycle 1 without DLT.
Measure: Number; unit: participants
Arm/Group | MLN0264 0.3 mg/kg | MLN0264 0.6 mg/kg | MLN0264 1.2 mg/kg | MLN0264 1.5 mg/kg | MLN0264 1.8 mg/kg | MLN0264 2.1 mg/kg | MLN0264 2.4 mg/kg
Number analyzed (Participants) | 2 | 2 | 2 | 2 | 6 | 4 | 1
participants | 0 | 0 | 0 | 0 | 1 | 2 | 1

2. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events and Serious Adverse Events
Description: An Adverse Event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (eg, a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug.
  A Serious Adverse Event (SAE) was any experience that suggests a significant hazard, contraindication, side effect or precaution that: results in death, is life-threatening, required in-patient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect or is medically significant.
  A treatment-emergent adverse event (TEAE) is defined as an adverse event with an onset that occurs after receiving study drug.
Time Frame: From the time informed consent is signed through 30 days after the last dose of study drug, approximately 9 months
Population: Safety Analysis Set included all participants who received at least one dose of study drug.
Measure: Number; unit: participants
Groups:
- MLN0264 Dose Escalation Phase: MLN0264 0.3 to 2.4 mg/kg, 30-minute intravenous (IV) infusion, Day 1 of each 21-day cycle, until disease progression or unacceptable toxicity or up to 1 year in the dose escalation phase.
Arm/Group | MLN0264 Dose Escalation Phase | MLN0264 1.8 mg/kg (mCRC Expansion)
Number analyzed (Participants) | 19 | 25
participants
  Adverse Events | 19 | 25
  Serious Adverse Events | 8 | 9

3. Primary Outcome: Maximum Tolerated Dose (MTD) of MLN0264
Description: MTD of MLN0264 was determined. Decisions regarding dose escalation were made based on any DLT that occurred during the first cycle of treatment.
Time Frame: Every 3 weeks until MTD is established, approximately 9 months
Population: as for outcome 1
Measure: Number; unit: mg/kg
Arm/Group | MLN0264 Dose Escalation Phase
Number analyzed (Participants) | 19
mg/kg | 1.8

4. Secondary Outcome: Best Overall Response
Description: The percentage of participants in each best overall response category, was determined using the Modified Response Evaluation Criteria in Solid Tumors (RECIST).
  Complete Response: Disappearance of all target lesions and all non-target lesions and normalization of tumor marker level.
  Partial Response: At least a 30% decrease in the sum of the Longest Diameter (LD) of target lesions, taking as reference the baseline sum LD.
  Progressive Disease (PD): At least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the start or the appearance of one or more new lesions. Appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions.
  Stable Disease: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD. Persistence of one or more non-target lesion(s) or/and maintenance of tumor marker level above the normal limits.
Time Frame: At the completion of every second cycle up to 12 cycles (approximately 9 months). Each cycle is a 21 days cycle
Population: Response Evaluable Population is defined as patients with measureable disease who receive any amount of MLN0264 and have at least 1 post-Baseline response assessment.
Measure: Number; unit: percentage of participants
Arm/Group | MLN0264 Dose Escalation Phase | MLN0264 1.8 mg/kg (mCRC Expansion)
Number analyzed (Participants) | 18 | 24
percentage of participants
  Complete Response (CR) | 0 | 0
  Partial Response (PR) | 6 | 0
  CR + PR | 6 | 0
  Stable Disease | 39 | 42
  Progressive Disease | 56 | 58

5. Secondary Outcome: Number of Participants With Antitherapeutic Antibodies (ATA)
Description: Blood was collected and sent to a laboratory to determine the immunogenicity, whether binding antibodies to MLN0264 were present (ATA development).
Time Frame: Day 1 of every 21 days cycle and at End of study (EOS) approximately 9 months
Measure: Number; unit: participants
Arm/Group | MLN0264 0.3 mg/kg | MLN0264 0.6 mg/kg | MLN0264 1.2 mg/kg | MLN0264 1.5 mg/kg | MLN0264 1.8 mg/kg | MLN0264 2.1 mg/kg | MLN0264 2.4 mg/kg | MLN0264 1.8 mg/kg (mCRC Expansion)
Number analyzed (Participants) | 2 | 2 | 2 | 2 | 6 | 4 | 1 | 25
participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

6. Primary Outcome: Cmax: Maximum Observed Serum Concentration for MLN0264
Description: Maximum observed serum concentration (Cmax) is the peak serum concentration of a drug after administration, obtained directly from the serum concentration-time curve. Cmax is reported for the 1.8 mg/kg dose, which is the MTD, where there is adequate data to provide robust parameter information reliably.
Time Frame: Cycle 1: Day 1 pre-dose to Day 21 post-dose
Population: Participants from the Pharmacokinetic (PK)-evaluable Population, all participants with sufficient dosing and reliable PK data to estimate PK parameters.
Measure: Geometric Mean (Full Range); unit: μg/mL
Arm/Group | MLN0264 1.8 mg/kg
Number analyzed (Participants) | 28
μg/mL | 48.63 [34.10 to 85.90]

7. Primary Outcome: Cmax: Maximum Observed Plasma Concentration for Monomethyl Auristatin E (MMAE)
Description: Maximum observed plasma concentration (Cmax) is the peak plasma concentration of a drug after administration, obtained directly from the plasma concentration-time curve. Cmax is reported for the 1.8 mg/kg dose, which is the MTD, where there is adequate data to provide robust parameter information reliably.
Time Frame: Cycle 1: Day 1 pre-dose to Day 21 post-dose
Population: as for outcome 6
Measure: Geometric Mean (Full Range); unit: ng/mL
Arm/Group | MLN0264 1.8 mg/kg
Number analyzed (Participants) | 28
ng/mL | 7.91 [4.02 to 18.10]

8. Primary Outcome: AUC0-21 Days: Area Under the Curve Day 0 to Day 21 for MLN0246
Description: Area under the drug concentration versus time curve from time 0 to Day 21. AUC0-21 is reported for the 1.8 mg/kg dose (the MTD), where there is adequate data to provide robust parameter information reliably.
Time Frame: Cycle 1: Day 1 pre-dose to 21 Days post-dose
Population: Participants from the PK-evaluable Population, all participants with sufficient dosing and reliable PK data to estimate PK parameters.
Measure: Geometric Mean (Full Range); unit: day*μg/mL
Arm/Group | MLN0264 1.8 mg/kg
Number analyzed (Participants) | 28
day*μg/mL | 67.81 [44.50 to 118.00]

9. Primary Outcome: AUC0-21 Days: Area Under the Curve Day 0 to Day 21 for MMAE
Description: Area under the plasma drug concentration versus time curve from time 0 to Day 21. AUC0-21 is reported for the 1.8 mg/kg dose (the MTD), where there is adequate data to provide robust parameter information reliably.
Time Frame: Cycle 1: Day 1 pre-dose to 21 Days post-dose
Population: Participants from the PK-evaluable Population, all participants with sufficient dosing and reliable PK data to estimate PK parameter AUC0-21 days.
Measure: Geometric Mean (Full Range); unit: day*ng/mL
Arm/Group | MLN0264 1.8 mg/kg
Number analyzed (Participants) | 26
day*ng/mL | 51.90 [24.50 to 150.00]

ADVERSE EVENTS:
Time Frame: From the time informed consent is signed through 30 days after the last dose of study drug (approximately 9 months)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | MLN0264 0.3 mg/kg | MLN0264 0.6 mg/kg | MLN0264 1.2 mg/kg | MLN0264 1.5 mg/kg | MLN0264 1.8 mg/kg | MLN0264 2.1 mg/kg | MLN0264 2.4 mg/kg
Serious Adverse Events (participants affected / at risk) | 0/2 | 2/2 | 1/2 | 0/2 | 10/28 | 2/4 | 1/1
Other Adverse Events (participants affected / at risk) | 2/2 | 2/2 | 2/2 | 2/2 | 28/28 | 4/4 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MLN0264 0.3 mg/kg (N=2) | MLN0264 0.6 mg/kg (N=2) | MLN0264 1.2 mg/kg (N=2) | MLN0264 1.5 mg/kg (N=2) | MLN0264 1.8 mg/kg (N=28) | MLN0264 2.1 mg/kg (N=4) | MLN0264 2.4 mg/kg (N=1)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 3 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Colonic obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Psoas abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Troponin T increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 — One treatment-emergent death occurred during the Dose Escalation Phase and is not related.
Convulsion (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MLN0264 0.3 mg/kg (N=2) | MLN0264 0.6 mg/kg (N=2) | MLN0264 1.2 mg/kg (N=2) | MLN0264 1.5 mg/kg (N=2) | MLN0264 1.8 mg/kg (N=28) | MLN0264 2.1 mg/kg (N=4) | MLN0264 2.4 mg/kg (N=1)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 | 10 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 4 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 7 | 3 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 5 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypothyroidism (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Periorbital oedema (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 7 | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 8 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 0 | 1 | 10 | 2 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 15 | 3 | 1
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 7 | 2 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 1 | 10 | 1 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chills (General disorders) | 0 | 1 | 0 | 0 | 2 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 0 | 0 | 13 | 1 | 1
Pain (General disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 0 | 10 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 6 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 8 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 0 | 0 | 3 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood magnesium decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Carbon dioxide increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 0 | 3 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 1 | 4 | 0 | 0
Liver function test abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 1 | 0 | 0 | 2 | 0 | 0
Mean cell haemoglobin concentration decreased (Investigations) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Mean cell volume decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Monocyte count decreased (Investigations) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Monocyte count increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neutrophil count increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 2 | 1 | 0
Platelet count increased (Investigations) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Transaminases increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 4 | 0 | 0
White blood cell count increased (Investigations) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 17 | 2 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 4 | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 2 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 5 | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 3 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 3 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 4 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 2 | 2 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 4 | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 2 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 4 | 0 | 1
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 5 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 3 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 4 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 9 | 1 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.